CLINICAL TRIAL: NCT06071208
Title: The National Plan To Prevent Diabetic Kidney Disease Among Egyptians: A Prospective Multicenter Randomized Controlled Study
Brief Title: Prevent Diabetic Kidney Disease Among Egyptians
Status: Not yet recruiting | Type: Observational
Sponsor: Fayoum University (Other)
Collaborators: Cairo University (Other); NewGiza University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine, Fayoum University
Other Study IDs: VCG 6
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus Without Complication
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases of study: Patients is diabetes whether recently discovered or long standing diabetes
  Interventions: Drug: Gliflozin
- controls of study: prediabetics ,or patients with clinical manifestations of insulin resistance eg acanthosis negricans
  Interventions: Drug: Gliflozin

INTERVENTIONS:
Drug: Gliflozin — to study whether the use of gliflozin prevented diabetic complications

SUMMARY:
Study of the possibility to prevent the development of Diabetic kidney disease in type 2 diabetic patients

DETAILED DESCRIPTION:
Study of the possible role of the SGLT2 inhibitors to prevent the development of frank type2 DM among prediabetic candidates.

Study of the possible role of the SGLT2 inhibitors to prevent the development of diabetic complications, namely diabetic kidney disease, diabetic retinopathy and neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* diabetics,prediabetics

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetics aged 18 years and above,male or females will be subjected to assessment of kidney functions at the beginning of the study and at the end to assess possibility of protective effect of SGLT-2,assessmentof other diabetic complications will be done also. Prediabetics will subjected to same assessment also
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-10-14 (Estimated); Primary Completion 2028-10-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
prevention of diabetic complications | 5 years
  glomerular filtration rate will be measured at the beginning of the study and at the end

CONTACTS AND LOCATIONS:
Overall Officials: Usama Sharaf El Din, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No